CLINICAL TRIAL: NCT04685317
Title: A Pilot Randomized Study of the Use of The Sentinel Device for Cerebral Protection During Atrial Fibrillation Ablation
Brief Title: Safety and Efficacy of the Sentinel Cerebral Protection Device in Atrial Fibrillation Ablation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Malini Madhavan (Other)
Responsible Party: Sponsor-Investigator, Malini Madhavan, Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 19-002836
Record Dates: First submitted 2020-12-22; First posted 2020-12-28 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Arrhythmia; Atrial Fibrillation
MeSH Terms: conditions — Arrhythmias, Cardiac; Atrial Fibrillation | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: Randomized study of Sentinel cerebral protection device vs no cerebral protection device in patients undergoing atrial fibrillation ablation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Sentinel® Cerebral Protection System Group (Experimental): Sentinel® Cerebral Protection System in patients undergoing AF catheter ablation
  Interventions: Device: Sentinel® Cerebral Protection System; Diagnostic Test: Magnetic Resonance Imaging
- Standard of Care Group (Active Comparator): Standard of care (no cerebral protection device) in patients undergoing AF catheter ablation
  Interventions: Diagnostic Test: Magnetic Resonance Imaging

INTERVENTIONS:
Device: Sentinel® Cerebral Protection System — A percutaneously delivered dual-filter protection device, designed to capture and remove debris dislodged during transcatheter aortic valve replacement procedures.
  Arms: Sentinel® Cerebral Protection System Group
Diagnostic Test: Magnetic Resonance Imaging — Cerebral MRI will be performed without gadolinium contrast using a 3 Tesla scanner prior to and 1 to 7 days after catheter ablation
  Other Names: MRI

SUMMARY:
The purpose of the study is to see if the Sentinel® Cerebral Protection System may prevent occurrence of stroke during an ablation procedure for atrial fibrillation (AF). The secondary purpose of this study is to study if cognitive function after AF ablation differs between those treated with the Sentinel cerebral protection device and those who do not receive the device.

DETAILED DESCRIPTION:
If assigned to receive the device, the Sentinel® Cerebral Protection System will be placed in your heart at the beginning of your ablation procedure, and then removed along with any collected blood debris upon completion of your procedure. The study team will then call you 30 days after your procedure to assess any neurological events. Your final visit will be 90 days after your procedure to complete a second 30 minute session of cognitive testing.

ELIGIBILITY:
Inclusion Criteria:

* Men / women over the age of 18 years undergoing radiofrequency, pulsed field or cryo-balloon ablation for AF in accordance with the current AHA/ACC/HRS guideline for management of patients with atrial fibrillation. This includes patients with symptomatic paroxysmal, persistent or long-standing persistent AF not responsive to or intolerant of a Class I or III anti-arrhythmic drug or patients with symptomatic paroxysmal or persistent AF prior to the initiation of a Class I or Class III antiarrhythmic drug). The decision to perform catheter ablation for AF will be made by the treating provider and the patient in accordance with the guidelines noted above. (January et al. J Am Coll Cardiol vol. 64, No. 21, 2014, page e1)
* Able to provide informed consent.
* Patients should have acceptable aortic arch anatomy and vessel diameters without significant stenosis as assessed using pre-procedure CT angiogram.

Exclusion Criteria:

* Anatomy unsuitable for use of Sentinel device:

  * Right extremity vasculature not suitable due to compromised arterial blood flow.
  * Brachiocephalic, left carotid or aortic arch not suitable due to excessive tortuosity, significant ectasia, stenosis (>70%), dissection or aneurysm.
* Cerebrovascular accident or transient ischemic attack within six months
* Carotid disease requiring treatment within six weeks
* Unable or unwilling to provide informed consent.
* Pregnant women
* Known history of dementia.
* Known hypersensitivity to nickel-titanium.
* Presence of MRI non-compatible implanted devices including cardiac implantable electronic devices.
* The presence of left atrial thrombus. All patients routinely undergo transesophageal echocardiogram prior to ablation and / or intra-cardiac echocardiogram at the beginning of the ablation procedure to rule out the presence of left atrial thrombus.
* Patients with a reversible cause for AF such as hyperthyroidism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incident of overt and covert CNS injury 7 days post AF ablation | 7 days post AF ablation
  Incidence of overt and covert CNS injury confirmed using physical examination and / or brain imaging during or within 7 days of the AF ablation
Incident of overt and covert CNS injury 90 days post AF ablation | 90 days post AF ablation
  Incidence of overt and covert CNS injury during or within 90 days of the AF ablation

SECONDARY OUTCOMES:
Change in neurocognitive function score | Baseline, 90 days
  Montreal cognitive assessment will administered at baseline and 90 days following ablation. Change in cognitive function score will be compared between the groups. The score ranges from 0 to 30 with higher score indicating better cognitive performance.
New cerebral infarcts | day 1 to 7 after atrial fibrillation ablation
  Total number of new cerebral infarcts in the protected territories detected on brain MRI after ablation in the Sentinel device group vs control group

CONTACTS AND LOCATIONS:
Overall Officials: Malini Madhavan, MBBS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials